CLINICAL TRIAL: NCT04995822
Title: Post Market Clinical Follow-up of EUROSTEM Femoral Stem
Status: Active, not recruiting | Type: Observational
Sponsor: EUROS (Industry)
Responsible Party: Sponsor
Other Study IDs: EC-309-01
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hip Osteoarthritis; Hip Arthropathy; Hip Arthritis; Hip Necrosis; Hip Fractures; Hip Dysplasia
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Fractures; Hip Dislocation | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EUROSTEM femoral stem: All patients who received EUROSTEM femoral stem whatever the version (cemented or cementless)
  Interventions: Device: hip arthroplasty

INTERVENTIONS:
Device: hip arthroplasty — Hip prosthesis surgery

SUMMARY:
EUROSSTEM is intended for use in primary and revision total hip replacement surgery.

Hip replacement is intended to provide increased patient mobility and reduce pain by replacing the damages hip joint articulation in patients where there is evidence of sufficient sound bone to seat and support the components.

As part of post market vigilance, EUROS will collect data on EUROSTEM performances and safety

DETAILED DESCRIPTION:
Post market observational study. This study is multicenter, prospective, non comparative.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received EUROSTEM
* Patient informed of its participation to the study
* Patient aged over 18 to date of surgery

Exclusion Criteria:

* Patient presenting a contraindication to EUROSTEM implantation.
* Patient who refused to participate to the study
* Vulnerable subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who fulfill the criteria of eligilibilty according to the instructions for use of EUROSTEM
Sampling Method: Non-Probability Sample
Enrollment: 131 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2032-11-06 (Estimated)

PRIMARY OUTCOMES:
Safety of EUROSTEM Femoral Stem | 1 year
  Collect the safety of the device trought complications occurence rate

SECONDARY OUTCOMES:
Radiological performances of EUROSTEM Femoral Stem | 1 year
  Collect the performances of the device trought radiological evaluation
Clinical performances of EUROSTEM Femoral Stem | 1 year
  Collect the performances of the device trought clinical scores
Survival of EUROSTEM Femoral Stem | 10 year
  Assess the survival rate of the device

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Clinique du Mail, Puilboreau, La Rochelle
  - Clinique Esquirol St Hilaire, Agen
  - CH Aix en Provence, Aix-en-Provence
  - Polyclinique du Beaujolais, Arnas
  - Clinique Montagard, Avignon
  - Polyclinique du Parc Drevon, Dijon
  - Clinique du Palais, Grasse
  - Hôpital privé Drôme Ardèche - Clinique Pasteur, Guilherand-Granges
  - Clinique Richelieu, Saintes

IPD SHARING:
Plan to Share IPD: No